CLINICAL TRIAL: NCT04751214
Title: Zaragoza Technique For Laparoscopic Appendicectomy
Brief Title: New Technique For Laparoscopic Appendicectomy
Status: Completed | Type: Observational
Sponsor: Israel De Alba Cruz (Other Government)
Responsible Party: Sponsor-Investigator, Israel De Alba Cruz, Principal Investigator, Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Organization: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Other Study IDs: IDC002
Record Dates: First submitted 2021-02-05; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Appendicitis Acute
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: APPENDICECTOMY

SUMMARY:
Introduction: Appendectomy is one of the most frequent emergency surgical procedures, currently with a preference for laparoscopic management worldwide. Objective: To report a new laparoscopic appendectomy technique and its results. Material and methods: study of patients with a diagnosis of appendicitis who are managed laparoscopically. In a total 1063 patients, 148 were operated on with the Zaragoza technique during the period from January 2002 to December 2018. The technique consists of making a window in the appendicular base between the meso and the appendicular wall, two prolene or silk sutures are placed, and the cecal appendix is cut between the two sutures, finally the mesoappendix is sectioned with a harmonic scalpel or bipolar clamp.

DETAILED DESCRIPTION:
this is a retrospective study based on files

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of appendicitis who are managed laparoscopically.

Exclusion Criteria:

* Less than 18 year old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: At the "General Ignacio Zaragoza" Regional Hospital, of the Institute of Social Security and Services for State Workers (ISSSTE), since July 2002, a new laparoscopic appendectomy technique has been performed by a surgical group.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2002-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
success of surgery | 2002-2018
  this study was revision of clinical files.
  measured by the rate of infection at the surgical site, mortality and hospital stay

IPD SHARING:
Plan to Share IPD: No